CLINICAL TRIAL: NCT07067138
Title: An Exploratory Study Using a Synthetic Lethality-Focused Algorithm to Identify Therapeutic Options in Advanced Metastatic Breast Cancer (SYNTHESIS-Breast)
Brief Title: A Synthetic Lethality-Focused Algorithm to Identify Therapeutic Options in Advanced Metastatic Breast Cancer (SYNTHESIS-Breast)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 10001891; 001891-C
Record Dates: First submitted 2025-07-12; First posted 2025-07-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-12

CONDITIONS: Breast Cancer; Breast Carcinoma; Cancer of the Breast; Malignant Neoplasm of Breast
Keywords: ENLIGHT; Triple Negative Breast Cancer (TNBC); Her2; NSR device
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1/No Recommended Match (Active Comparator): Treatment per physician's choice
  Interventions: Device: Expression Networks for highLIGHting Tumor vulnerabilities (ENLIGHT); Device: TruSight(R) Oncology 500; Device: TruSeq Matched Tumor Normal Whole Exome Sequencing Assay
- 2/Genomic Marker Associated with FDA-Approved On-Label Treatment (Experimental): Treatment in accordance with genomic marker; treatment to be directed locally by referring/treating physician
  Interventions: Device: Expression Networks for highLIGHting Tumor vulnerabilities (ENLIGHT); Device: TruSight(R) Oncology 500; Device: TruSeq Matched Tumor Normal Whole Exome Sequencing Assay
- 3/Transcriptomic Match (Experimental): Treatment regimen as selected by transcriptomic algorithm; treatment to be directed by NIH study team with requirement for treatment at NIH
  Interventions: Device: Expression Networks for highLIGHting Tumor vulnerabilities (ENLIGHT); Device: TruSight(R) Oncology 500; Device: TruSeq Matched Tumor Normal Whole Exome Sequencing Assay

INTERVENTIONS:
Device: Expression Networks for highLIGHting Tumor vulnerabilities (ENLIGHT) — This is a computational algorithm that takes RNA-seq data from tumor FFPE blocks and, given a list of pre-specified treatments, generates as output the predicted responses to those treatments.
Device: TruSight(R) Oncology 500 — TSO500 uses formalin-fixed, paraffin-embedded (FFPE) tumor blocks to generate a 523-gene DNA panel (with tumor mutational burden and microsatellite instability) to assess for biomarkers linked to FDA-approved, on-label therapies as well as whole-exome RNA-seq that can be used with the ENLIGHT algorithm.
Device: TruSeq Matched Tumor Normal Whole Exome Sequencing Assay — The TruSeq Matched Tumor-Normal Whole Exome Sequencing assay is a next-generation sequencing assay that uses tumor DNA from formalin-fixed, paraffin-embedded (FFPE) tumor blocks and germline DNA drawn from blood to provide extended sequencing information on the tumor as well as any pathogenic variants, likely pathogenic variants, and variants of uncertain significance in 156 genes from the normal blood sample.

SUMMARY:
Background:

Breast cancer is the most common cancer in US women. There are different types of breast cancers; some are aggressive and difficult to treat. Researchers want to know if an algorithm (ENLIGHT) can help choose approved drugs that will treat these cancers more effectively.

Objective:

To test whether ENLIGHT can find better treatments for aggressive breast cancers.

Eligibility:

People aged 18 years and older with triple-negative or endocrine therapy resistant breast cancer; the cancer must have either failed to respond to treatment or come back after treatment.

Design:

Participants will be screened. A sample of tissue taken from the tumor will be tested using ENLIGHT as well as another method (TruSight Oncology 500).

Participants will be assigned to 1 of 3 groups based on the algorithm search results:

Group 1: No drug option was recommended. Participants will continue with their standard treatment with their local doctors.

Group 2: A drug already approved for the participant's disease was recommended, but the participant has not yet received it. These results will be sent to the participant's local doctors. Participants may return to the NIH if their disease gets worse after using the suggested drugs.

Group 3: A drug approved for other uses was recommended. Participants will be treated with the recommended drugs at the NIH; their care will be managed by an NIH doctor. They will continue to receive treatment as long as the drugs are helping them. They will have follow-up visits for 2 years after treatment ends.

Participants who are not treated at the NIH will be contacted for a check on their health every 3 months for 2 years.

DETAILED DESCRIPTION:
Background:

* While 10-20% of breast cancers diagnosed in the U.S. are "triple-negative" (TNBC), the 5-year survival rate among TNBC patients with metastatic disease at diagnosis is 12%, and median survival after recurrence is approximately 24 months, demonstrating clear need for additional therapeutic options.
* Patients with metastatic hormone-receptor positive (HR+) breast cancer who develop endocrine-refractory disease (that is, no longer responsive to combinations including endocrine therapy) also suffer from a dearth of therapeutic options beyond cytotoxic chemotherapy, with overall survival after standard of care treatment (as seen across recent trials) often less than 1 year.
* Personalized oncology strategies have the potential to identify therapies across multiple cancer types. However, such strategies (which currently use patient DNA sequencing) only select a small subgroup of candidate patients by targeting direct matches in their cancers necessitating approaches that can broaden the pool of patients who may benefit from targeted therapies.
* Recent computational approaches are able to leverage additional -omics data, such as whole-transcriptome RNA-seq, and relationships between genes, such as synthetic lethality, to better predict responses to off-label targeted therapy or immunotherapy treatments compared to single-target strategies in retrospective clinical trial data.
* This study will apply the use of one such published computational transcriptomics algorithm, ENLIGHT, to prospectively identify therapeutic options for participants with metastatic breast cancer who currently experience limited treatment options.

Objectives:

* Part A: To assess the feasibility of using the ENLIGHT algorithm to match heavily pretreated participants with metastatic breast cancer to off-label therapies
* Part B (If feasibility-run in is met): To assess the objective response rate (ORR) of participants with advanced breast cancer using treatment recommended by the computational transcriptomics algorithm ENLIGHT

Eligibility:

* Participants must have a histologically confirmed diagnosis of metastatic breast cancer.
* Participant tumor subtypes will be enrolled as follows:

  * TNBC Cohort: TNBC will be defined as estrogen receptor (ER) < 10% or progesterone receptor (PR) <10% by immunohistochemistry (IHC).
  * Endocrine-Refractory Cohort: HR+ (ER positive and/or PR positive). HR+ will be defined as ER >=10% or PR >= 10% by IHC.
  * For both cohorts, HER2 will be considered negative if not amplified as per ASCO-CAP guidelines per IHC/FISH. Note: HER2-low status will be regarded in accordance with NCCN guidelines (in which this designation serves as a predictive marker for trastuzumab deruxtecan, but participants are otherwise not considered eligible for other HER2-directed therapies).
* Participants must have been treated with at least one line of standard systemic therapy after diagnosis of metastatic disease, have progressive disease on their current regimen, and must not be eligible for another approved/standard therapy that has been shown to improve overall survival.
* Participants with HR+ disease must be deemed refractory to endocrine therapy per their clinical team, with concordance by study team.
* Participants must have measurable disease per RECIST v1.1.
* Archival tumor (preserved via FFPE) must be available from a biopsy performed within the past 6 months, or participants will need to undergo core biopsy and have at least one amenable tumor for the procedure, to optimize reliability of ENLIGHT results.
* Age >=18 years

Design:

* This is an exploratory study that uses the ENLIGHT algorithm (Pangea Biomed) on whole-exome RNA-seq extracted from FFPE tissue to recommend and prioritize off-label therapies for participants.
* FFPE blocks from biopsies performed locally may be submitted if obtained 6 months or less prior to study enrollment, or biopsies may be obtained at the NIH in those participants for whom archival tissue is not available and there is at least one measurable site of disease that is deemed safe to biopsy.
* All RNA-seq extraction and sequencing will be performed by the CLIA-certified Laboratory of Pathology at the Center for Cancer Research, National Cancer Institute.
* Using the ENLIGHT algorithm to recommend and prioritize possible treatment options will test utility of this algorithm, which leverages RNA-seq, to add to clinical decision support.
* While on treatment at the NIH, participants will be asked to provide both blood correlative samples and an optional post-treatment tissue biopsy at day 15 / start of cycle 2 as per their treatment protocol.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Participants must have a histologically confirmed diagnosis of metastatic breast cancer. Note: Pathology testing outside NIH will be accepted for eligibility purposes.
2. Participant tumor subtypes will be enrolled as follows:

   * TNBC Cohort: TNBC will be defined as ER < 10% or PR < 10% by immunohistochemistry (IHC).
   * Endocrine-Refractory Cohort: HR+ (ER+ and/or PR+) will be defined as ER >= 10% or PR >= 10% by IHC.
   * For both cohorts, HER2 will be considered negative if not amplified as per ASCOCAP guidelines per IHC/FISH. Note: HER2-low status will be regarded in accordance with NCCN guidelines (in which this designation serves as a predictive marker for trastuzumab deruxtecan, but participants are otherwise not considered eligible for other HER2-directed therapies).
3. Participants must have been treated with at least one (1) line of systemic therapy after diagnosis of metastatic disease, have progressive disease or adverse events requiring discontinuation of their current regimen, and must not be able to transition to another approved systemic therapy shown to improve overall survival.

   -Participants with HR+ disease must be deemed refractory to endocrine therapy per their clinical team, with concordance by study team.

   Note: Participants who cannot receive standard therapy that has been shown to prolong overall survival due to concurrent medical issues versus progression of disease will be eligible, if other eligibility criteria are met. If appropriate, participants may remain on treatment during biopsy, screening and initial tissue review/testing for this study. However, their clinical team must confirm that the current line of treatment no longer offers benefit prior to the time of reporting and treatment assignment.
4. Participants must have measurable disease per RECIST v1.1. Note: Palliative radiotherapy to site(s) of disease may be completed during screening as long as disease outside of the planned sites of radiation is available for response assessment.
5. Archival tumor (preserved via FFPE) must be available from a biopsy performed within the past 6 months. The timeframe of 6 months is required to optimize reliability of ENLIGHT results. It is assumed that a participant has had no more than one (1) line of systemic treatment since the last biopsy. Participants who have had multiple intervening lines of therapy since biopsy was obtained will be reviewed by the study team to determine if another biopsy may be needed. Note: If archival tissue is not available within that timeframe, tissue from the next scheduled biopsy can be sent to NIH for testing. If it is not possible for a biopsy to be scheduled, the study team will evaluate the possibility of a biopsy being performed at the NIH for enrollment purposes.
6. Age >=18 years.
7. ECOG performance status <2 (Karnofsky >60%)
8. Participants must have organ and marrow function as defined below:

   * Leukocytes >= 3,000/mcL
   * Hemoglobin >= 8g/dL
   * Absolute neutrophil count >= 1,200/mcL
   * Platelets >=75,000/mcL
   * Total bilirubin <= 1.5 x institutional upper limit of normal (In the case of known Gilbert's Disease, total bili >1.5 may be considered.)
   * AST(SGOT)/ALT(SGPT) <= 3x institutional upper limit of normal
   * Creatinine < 1.5 x normal institutional limits OR Creatinine clearance >=60 mL/min/1.73 m2
9. Ability to take oral medications.
10. Participants with an existing diagnosis of diabetes or hypertension, must have disease well-controlled with at least annual physician follow-up.
11. Women of child-bearing potential and men with a partner of child-bearing potential must be willing to use appropriate contraception in the event that they match to a therapy that requires such. The duration of contraception use will depend on the therapy assigned.
12. Willingness to comply with required study procedures and visits for the duration of study.
13. Participants with asymptomatic brain metastases may be included if metastases have been previously treated with local therapy including radiation at least 4 weeks prior to first dose of treatment and there is no indication for additional local therapy (including active progression).
14. Participants with human immunodeficiency virus (HIV) must be on an effective antiretroviral therapy with undetectable viral load for at least the last 6 months.
15. Participants with evidence of chronic hepatitis B virus (HBV) infection, must have HBV viral load that is undetectable on suppressive therapy, if indicated.
16. Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection must be currently on treatment, with undetectable HCV viral load.
17. Participants with a prior or concurrent malignancy are eligible if the natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the off-label therapies offered on this study in the opinion of the Principal Investigator (PI) and are otherwise eligible for this trial.
18. Participants with current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. Note: To be eligible for this trial, participants should be class 2B or better.
19. Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Participants in active visceral crisis, symptomatic brain metastases requiring local therapy, or active leptomeningeal disease given the time required for testing and therapy selection.
2. Participants with uncontrolled intercurrent illness evaluated by physical exam and chemistries or situations that would limit compliance with study requirements, interpretation of results or that could increase risk to the participant.
3. Participants with the following active cardiac conditions: symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia (per medical record).
4. Participants with lung disease requiring continuous oxygen supplementation.
5. Participants with decompensated cirrhosis and/or end-stage kidney disease on dialysis.
6. Participants with positive serum or urine beta-HCG pregnancy test performed at screening.
7. Participants who are unable to provide tissue specimens of sufficient quality for use in this study. Quality of DNA and RNA is determined during screening. This may be due to issues with biopsy sample collection, inadequate RNA extraction, or quality control failure. Participants may be re-screened if initial specimens are not adequate, if they are amenable to re-biopsy, and additional site(s) of disease for adequate re-sampling are available.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-08-04 (Estimated); Study Completion 2029-08-04 (Estimated)

PRIMARY OUTCOMES:
Part A: To assess the feasibility of using the ENLIGHT algorithm to match heavily pretreated participants with metastatic breast cancer to off-label therapies | Assessed after the Reporting Visit of the 20th participant to the study, and to be completed before Part B
  The number of participants of the first 20 enrolled overall having a match via ENLIGHT and being assigned to Arm 3.
Part B: (If feasibility lead-in met) To assess the objective response rate (ORR) of participants with advanced breast cancer using treatment recommended by the ENLIGHT algorithm | Every 2 cycles until progression of disease, completion of treatment, or 2 years after treatment initiation (whichever comes first)
  ORR is reported as a single endpoint measure (percentage) at time of interim analysis and at time of study completion and will be accompanied by a 95% confidence interval.

SECONDARY OUTCOMES:
To determine the overall frequency of the ENLIGHT algorithm in recommending matches of targeted therapy or immunotherapy for participants who would otherwise be ineligible per existing biomarkers associated with FDA-approved, on-label treatments | Every 2 cycles until progression of disease, completion of treatment, or 2 years after treatment initiation (whichever comes first)
  Fraction of the eligible participants who match with a treatment by ENLIGHT along with a 95% confidence interval on the fraction, separately by cohort
To assess the duration of clinical benefit for treatments recommended by the ENLIGHT algorithm | Every 2 cycles until progression of disease, completion of treatment, or 2 years after treatment initiation (whichever comes first)
  Reported using the Kaplan-Meier method along with the median duration of clinical benefit and its 95% confidence interval, separately by cohort
To determine the specific agents for which ENLIGHT demonstrates the best predictive performance in the context of breast cancer | Ongoing
  Frequency of patients matched to therapeutic options on study (Count of participants per unique therapy in Arm 3)
To determine extent of therapy associated toxicity burden and related outcomes for participants who are matched to a therapy through the ENLIGHT algorithm | At least Day 1 of each cycle, throughout treatment, and at the end-of treatment visit; then every 3 months for up to 2 years.
  Frequency of adverse events (AE) per CTCAE v5.0, by type and grade of toxicity
To assess the ORR/duration of clinical benefit for participants undergoing an additional iteration of treatment as recommended by the ENLIGHT algorithm | Every 2 cycles until progression of disease, completion of treatment, or 2 years after treatment initiation (whichever comes first)
  Reported using the Kaplan-Meier method along with the median duration of clinical benefit and its 95% confidence interval, separately by cohort

CONTACTS AND LOCATIONS:
Overall Officials: Padma S Rajagopal, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication. Data not published in a manuscript will be shared via public source once the data set completes QC. Clinical data will be made available during the study and indefinitely via BTRIS.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians. Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001891-C.html